CLINICAL TRIAL: NCT02070705
Title: The Use of Dynamic Contrast Enhanced Magnetic Resonance Imaging (DCE MRI) in the Management of Pancreatic Cancer
Brief Title: DCE MRI in Patients With Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Oregon Health and Science University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alexander Guimaraes, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00009694; NCI-2014-00270 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MR00045736; CR00022704; IRB00009694 (Other: OHSU Knight Cancer Institute); K08EB012859 (NIH); U01CA278923 (NIH)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Familial Pancreatic Cancer; Pancreatic Adenocarcinoma; Pancreatic Intraductal Papillary-Mucinous Neoplasm
MeSH Terms: conditions — Pancreatic carcinoma, familial; Pancreatic Intraductal Neoplasms | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (High-risk for familial/hereditary pancreatic cancer) (Experimental): Patients undergo DCE MRI (Dynamic Contrast-Enhanced Magnetic Resonance Imaging with Ferumoxytol) yearly for a minimum of 3 scans.
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Drug: Ferumoxytol
- Arm II (IPMN) (Experimental): Patients undergo DCE MRI (Dynamic Contrast-Enhanced Magnetic Resonance Imaging with Ferumoxytol) prior to surgery for resection of IPMN.
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Drug: Ferumoxytol
- Arm III (Pancreatic cancer) (Experimental): Patients who undergo chemotherapy prior to resection will have 2 DCE MRI scans; one study scan prior to undergoing neoadjuvant therapy, as well as one study scan following neoadjuvant therapy as part of their pre-operative work up in addition to the standard imaging studies. For patients that do not require chemotherapy treatment prior to resection they will have just one DCE MRI scan prior to surgical resection. Patients currently undergoing neoadjuvant therapy or who have already completed neoadjuvant therapy that were unable to undergo imaging at baseline and are now proceeding to resection will have one DCE MRI scan prior to surgical resection.
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Drug: Ferumoxytol
- Arm IV (Healthy volunteers) (Active Comparator): Patients undergo a single DCE MRI (Dynamic Contrast-Enhanced Magnetic Resonance Imaging with Ferumoxytol) examination.
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Drug: Ferumoxytol

INTERVENTIONS:
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo DCE MRI
  Other Names: DCE; DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; Ferumoxytol Non-Stoichiometric Magnetite

SUMMARY:
This clinical trial studies an imaging technique known as dynamic contrast enhanced magnetic resonance imaging (DCE MRI) in identifying the presence of pancreatic cancer. DCE MRI is a procedure that takes detailed pictures of functional and structural properties inside the body using magnetic field imaging. These images may better characterize pancreatic cancer in patients at high risk or in patients who may have undergone chemotherapy for pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the ability of DCE-MRI to identify the presence of pancreatic cancer in patients at high risk for hereditary pancreatic cancer.

II. Assess the ability of DCE-MRI to identify the presence of pancreatic cancer in patients with cystic lesions of the pancreas.

III. Assess the ability of DCE-MRI to accurately predict tumor margins in patients who have undergone chemotherapy for pancreatic cancer.

IV. Obtain DCE-MRI scans of from healthy volunteers (Group 4), to establish baseline imaging parameters of the normal, non-diseased pancreas for use as a comparator to affected pancreata.

SECONDARY OBJECTIVE:

I. Clinical factors associated with the presence of pancreatic cancer will be assessed in each of the three experimental groups, including disease free survival and overall survival.

II. Additional MRI pulses sequences (e.g. MR fingerprinting, etc.) will be acquired for the assessment of tissue contrast before and after the administration of contrast agents.

OUTLINE: Patients are assigned to 1 of 4 groups.

ARM I (High-risk for familial or hereditary pancreatic cancer): Patients undergo DCE MRI yearly for a minimum of 3 scans.

ARM II (Intraductal papillary mucinous neoplasms [IPMN]): Patients undergo DCE MRI prior to surgery for resection of IPMN.

ARM III (Pancreatic cancer): Patients who undergo chemotherapy prior to resection will have 2 DCE MRI scans; one study scan prior to undergoing neoadjuvant therapy, as well as one study scan following neoadjuvant therapy as part of their pre-operative work up in addition to the standard imaging studies. For patients that do not require chemotherapy treatment prior to resection they will have just one DCE MRI scan prior to surgical resection. Patients currently undergoing neoadjuvant therapy or who have already completed neoadjuvant therapy that were unable to undergo imaging at baseline and are now proceeding to resection will have one DCE MRI scan prior to surgical resection.

ARM IV (Healthy volunteers): Patients undergo a single DCE MRI examination.

ELIGIBILITY:
Inclusion Criteria:

* ALL PARTICIPANTS: A negative serum or urine pregnancy test for woman of childbearing potential
* ALL PARTICIPANTS: Ability to understand and the willingness to sign a written informed consent document
* GROUPS 1, 2, AND 3: "All participants" described above
* GROUPS 1, 2, AND 3: Must be consented for the Oregon Pancreatic Tumor Registry (OPTR)
* GROUPS 1, 2, AND 3: Group 1: participants identified as being high-risk for familial or hereditary pancreatic cancer, and must conform to one or more of the following requirements:

  * Have a strong family history of pancreatic cancer; this is defined as pancreatic cancer occurring in one first- degree relative and two other relatives, or two first- degree relatives; or,
  * Have a known high-risk genetic syndrome (e.g., BRCA 1&2, STK11, CDNK2A, PRSS1, and MSH 2&6)
* GROUPS 1, 2, AND 3: Group 2 participants identified as having IPMN on standard radiographic imaging that meets criteria for resection based on symptoms or on conventional imaging (computed tomography [CT] or MRI) findings
* GROUPS 1, 2, AND 3: Group 3 participants must have pathologically- confirmed pancreatic adenocarcinoma, with or without the need for neoadjuvant chemotherapy prior to surgical resection.
* HEALTHY VOLUNTEERS (Group 4): Must meet inclusion criteria for "all participants" described above
* HEALTHY VOLUNTEERS (Group 4): Group 4 participants must have no history of cancer, pancreatic disease, or family history of pancreatic cancer.

  * Family history will be defined as pancreatic cancer occurring in one first-degree relative and two other relatives, or two first-degree relatives

Exclusion Criteria:

* Participants unable or unwilling to give written, informed consent or to undergo MRI imaging
* Participants with multiple drug allergies, and/or subjects who have had an allergic reaction to any intravenous iron replacement product, or a known history of hypersensitivity to ferumoxytol
* Participants with concurrent clinical diagnosis, evidence of suspected hemochromatosis, or other diseases of iron metabolism (i.e., iron overload)
* Cirrhosis, cardiomyopathy, restrictive heart disease, or bronzing of the skin
* Pregnant women are excluded from this study because there is an unknown, but potential risk, for adverse events, as small animal trials have linked ferumoxytol administration (at very high doses) to birth defects (e.g., soft-tissue malformations and decreased fetal weights); it is not known whether ferumoxytol is present in human milk; breastfeeding, however, should be discontinued if the mother receives ferumoxytol while nursing
* Human immunodeficiency virus (HIV)-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ferumoxytol
* Participants with diagnosis of renal insufficiency or glomerular filtration rate (GFR) < 60 ml/min/1.73m^2
* Adult patients who require monitored anesthesia for MRI scanning
* Participants with any contraindications to gadolinium-based contrast agents
* Participants who have a contraindication for MRI (e.g. metal in their bodies, a cardiac pacemaker, or other incompatible device), or are severely agitated or claustrophobic. (For patients that are eligible but there is a concern of metal in their bodies, the will be given the option if interested to have a x-ray completed prior to study enrollment to determine if they can proceed with the study MRI. Patients with a concern of metal in their bodies that don't agree to a x-ray will not be enrolled into the study.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Presence of pancreatic cancer (yes or no) for patients that are either at high risk for hereditary pancreatic cancer (Group I) | Up to 5 years
  Descriptive statistical analysis will be conducted for primary endpoints.
Presence of pancreatic cancer (yes or no) for patients with cystic lesions of the pancreas (Group II) | Up to 5 years
  Descriptive statistical analysis will be conducted for primary endpoints.
Change in tumor margins in patients who have undergone chemotherapy for pancreatic cancer (Group III) | Baseline to up to 2 years
  The change of dynamic contrast enhanced magnetic resonance imaging (DCE MRI) parameters from baseline will be correlated with the tumor margins determined by pathological specimen following surgical resection through linear regression model.

SECONDARY OUTCOMES:
Disease free survival (Group I) | Time of enrollment to time of diagnosis, assessed up to 5 years
  Kaplan-Meier method will be used to estimate the survival distribution for disease free survival. The estimated median and 95% confidence interval will be computed.
Disease free survival (Group II) | Time of surgical resection to time of disease recurrence, if applicable, assessed up to 5 years
  Kaplan-Meier method will be used to estimate the survival distribution for disease free survival. The estimated median and 95% confidence interval will be computed.
Disease free survival (Group III) | Time of surgical resection to time of recurrence, assessed up to 5 years
  Kaplan-Meier method will be used to estimate the survival distribution for disease free survival. The estimated median and 95% confidence interval will be computed.
Overall survival (Group I) | Time of surgical resection to time of death, assessed up to 5 years
  Kaplan-Meier method will be used to estimate the survival distribution for overall survival. The estimated median and 95% confidence interval will be computed.
Overall survival (Group II) | Time of surgical resection to time of death, assessed up to 5 years
  Kaplan-Meier method will be used to estimate the survival distribution for overall survival. The estimated median and 95% confidence interval will be computed.
Overall survival (Group III) | Time of surgical resection to time of death, assessed up to 5 years
  Kaplan-Meier method will be used to estimate the survival distribution for overall survival. The estimated median and 95% confidence interval will be computed.
Surgical pathological diagnosis and T & N stage according to the American Joint Committee on Cancer (AJCC) tumor, node, metastasis (TNM) staging system (Group II) | At time of surgery
  Will be assessed as potential confounders or effect modifiers in the model. Will report c-statistics for each model.
Surgical pathological diagnosis and T & N stage according to the AJCC TNM staging system (Group III) | At time of surgery
  Will be assessed as potential confounders or effect modifiers in the model. Will report c-statistics for each model.
Resection margin status (R0, R1 or R2) (Group III) | At time of surgery
  Will be assessed as potential confounders or effect modifiers in the model. Will report c-statistics for each model.
DCE- MRI imaging parameters (Group I) | Up to 5 years
  The DCE- MRI parameters will be obtained from the pancreases in the control group and will be descriptively analyzed for use as a comparison in other groups.
DCE- MRI imaging parameters (Group II) | Once prior to surgery
  The DCE- MRI parameters will be obtained from the pancreases in the control group and will be descriptively analyzed for use as a comparison in other groups.
DCE- MRI imaging parameters (Group III) | Up to 5 years
  The DCE- MRI parameters will be obtained from the pancreases in the control group and will be descriptively analyzed for use as a comparison in other groups.
DCE- MRI imaging parameters and descriptional analysis of normal pancreas DCE- MRI images (Group IV) | Once at time of enrollment
  The DCE- MRI parameters will be obtained from the pancreases in the control group and will be descriptively analyzed for use as a comparison in other groups.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Guimaraes, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States